CLINICAL TRIAL: NCT02915419
Title: Evaluation of Survival of Mature Second Premolar With Periapical Lesion Following Different Regenerative Treatment Protocols
Brief Title: Evaluation of Survival of Mature Second Premolar Treated With Regenerative Techniques
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Wagih Tarek Ali, assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEBD-CU-2016-09-203
Record Dates: First submitted 2016-09-20; First posted 2016-09-27 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Carious Teeth
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- group A (Active Comparator): prp revascularization
  Interventions: Biological: PRP; Biological: PRF
- group B (Experimental): treatment of affected teeth using platelet rich fibrin by applying prf in steril root canal
  Interventions: Biological: PRP; Biological: PRF

INTERVENTIONS:
Biological: PRP — platelet rich plasma
Biological: PRF — PLATELET RICH FIBRIN

SUMMARY:
This study aims to compare the ability of different regenerative protocols in the treatment of mature necrotic

DETAILED DESCRIPTION:
American Dental Association adopted the tissue engineering concept and pulp regeneration in 2009. Regeneration was focused on the treatment of immature necrotic teeth so as to allow root completion, improving both the functionality and durability of the affected tooth. Utilizing a blood clot in the affected tooth with immature roots was very beneficial, as it acts as a scaffold for the migration of stem cells and morphogens to allow regeneration .

Based on the success of pulp regeneration in treating immature teeth, ambitious dentists started to look forward on regenerating the pulp of mature teeth as a substitution to the conventional root canal treatment. On the other hand, lots of clinicians were very doubtful about treating mature teeth with the same protocol, as the small apical foramen might not provide a good portal for the entry of stem cells and growth factors, which in turn is very important for the success of pulp regeneration.Doubts in treating mature apex encouraged researchers to look for an alternative to the stem cells other than the apical papilla, from this concept the idea for using an alternative source of stem cells and growth factors as platelet rich plasma (PRP) emerged. The use of platelet rich plasma (PRP) as a potentially ideal scaffold for regenerative endodontic therapy has been reported in the treatment of immature teeth. However, the use of bovine thrombin for the activation of PRP has been an issue of controversy, as it requires non autologous anticoagulant known to hinder the process of pulp regeneration.

This led to the development of the second generation, platelet concentrate known as Choukroun's platelet rich fibrin (PRF) which is totally autologous in nature. Platelet rich fibrin (PRF) was very promising, but it is debatable whether to use PRP or PRF.The objective of this study is to evaluate novel regenerative techniques, utilizing platelet rich plasma and platelet rich fibrin in treatment of second premolar teeth with necrotic pulp, mature apex, and periapical lesion. This is a trial to prolong the survival of the affected tooth, and to aid in complete healing of periapical lesion, and to regain pulp vitality and sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are free from any physical or mental handicapping condition with no underlying systemic diseases.

Non-pregnant females Single canalled second premolar

* Patients having non-vital, mature, second premolar teeth, radiographic evidence of periapical lesion.
* Positive patient/Guardian compliance for participation in the study.

Exclusion Criteria:

* Any known sensitivity or adverse reactions to medicaments or pharmaceuticals necessary to complete the trial.

Non-restorable coronal portion of teeth involved in the trial. Vital teeth Immature teeth Traumatized teeth Radiographic evidence of external or internal root resorption. Any criterion, not mentioned in the inclusion criteria

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Survival | 1 year
  how long will the tooth survive after treatment, testing the durability of tooth

SECONDARY OUTCOMES:
healing | 1 year
  measuring the density of lesion using the cone beam CT
vitality | 1 year
  after how many days will the tooth respond normaly to stimulus

OTHER OUTCOMES:
sensitivity | 1 year
  after how many days will the tooth respond positively to electric pulp tester

CONTACTS AND LOCATIONS:
Overall Officials: wagih ali, ass lecturer, Principal Investigator — Cairo University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wang Y, Zhu X, Zhang C. Pulp Revascularization on Permanent Teeth with Open Apices in a Middle-aged Patient. J Endod. 2015 Sep;41(9):1571-5. doi: 10.1016/j.joen.2015.04.022. Epub 2015 Jun 10. PMID 26071100